CLINICAL TRIAL: NCT01280669
Title: Sirolimus as a Therapeutic Approach for Uveitis: A Phase 2, Open-label, Randomized Study to Assess the Safety, Tolerability, and Bioactivity of Two Doses of Intravitreal Injection of Sirolimus in Patients With Non-infectious Uveitis
Brief Title: Intravitreal Sirolimus as Therapeutic Approach to Uveitis
Acronym: SAVE-2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Never started due to sponsor decision
Sponsor: Stanford University (Other)
Collaborators: Santen Inc. (Industry)
Responsible Party: Principal Investigator, Quan Dong Nguyen, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00046190
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Uveitis; Intermediate Uveitis; Posterior Uveitis; Panuveitis
Keywords: Non-infectious; Uveitis; Panuveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Uveitis, Posterior; Panuveitis | interventions — Intravitreal Injections; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Intravitreal injections of 440mcg sirolimus (low-dose monthly group)
  Interventions: Drug: Intravitreal injection 440mcg
- Group 2 (Experimental): Intravitreal injections of 880mcg sirolimus (high-dose every other month group)
  Interventions: Drug: Intravitreal injection of sirolimus 880mcg

INTERVENTIONS:
Drug: Intravitreal injection 440mcg — Intravitreal injections of sirolimus 440mcg/20mcL at baseline and months 1, 2, 3, 4, and 5.
  Other Names: Low-dose; Monthly
  Arms: Group 1
Drug: Intravitreal injection of sirolimus 880mcg — Intravitreal injection of 880mcg/20mcL sirolimus at baseline and months 2 and 4.
  Other Names: High-dose; Bi-monthly
  Arms: Group 2

SUMMARY:
The purpose of this study is to find out about the safety and effectiveness of two different doses the study drug, sirolimus, administered intravitreally in patients with uveitis. The potential effectiveness of sirolimus can be utilized to control inflammation in uveitis and yet avoid the potential complications that are usually associated with the systemic use of the drug and other immunomodulatory therapies. In this study, the investigators will administer sirolimus inside the eye (intravitreally) in one of two doses (440mcg/mcL or 880mcg/mcL). Local administration of sirolimus to the eye is not expected to have effects on the rest of the body. Therefore, it may offer a safer way than the current methods used to control the inflammation caused by non-infectious uveitis.

DETAILED DESCRIPTION:
Uveitis is a condition in which certain parts of your eye become inflamed. The inflammation is usually recurrent. If the inflammation is not treated adequately, permanent damage to the eye and to the vision may occur. The inflammation can be caused by infectious or non infectious causes. The current research is being done to determine the safety and the usefulness of treatment of non-infectious uveitis using different doses of intravitreal injections of a drug called sirolimus.

Current treatment options for uveitis include oral corticosteroids and drugs that weaken the immune system of the body (i.e., immunosuppressant drugs). Treatment using oral corticosteroids, especially for long periods, may cause many undesirable side effects and complications such as high blood sugar, high blood pressure, bone weakness, obesity, stomach ulcers, abnormal hair growth, and increased risks of infection. In addition to that, in some cases, the disease cannot be controlled even with the highest dose of steroids.

Injection of steroids around and inside the eye can be used to control uveitis. However, the inflammation does not always respond to such kind of treatment. The eyes may develop high pressure and cataract with injections of steroids into the eyes or around the eyes.

On the other hand, despite their potential effectiveness, treatment with drugs that weaken the immune system may cause severe side effects. Increased risk of infection is a common side effect of all the immunosuppressant drugs. The immune system protects the body from infections. When the immune system is suppressed, infections are more likely to happen. Some of these infections are potentially dangerous. Because the immune system protects the body against some forms of cancer, immunosuppressant drugs are also associated with a slightly increased risk of cancer. For example, long-term use of immunosuppressant drugs may carry an increased risk of developing skin cancer as a result of the combination of the drugs and exposure to sunlight. The immunosuppressive drugs are very powerful and can cause serious side effects such as high blood pressure, kidney problems, and liver problems. Some side effects may not show up until years after the medicine is used.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females greater than or equal to 12 years of age.
2. Able to give informed consent and attend all study visits.
3. Have diagnosis of uveitis determined by the Investigator to be non-infectious based on the patient's medical history, history of present illness, ocular examination, review of systems, physical examination, and any pertinent laboratory evaluations.
4. Meet the following criteria:

   * Have active uveitis, defined as having at least 1+ Vitreous Haze and/or at least 1+ Vitreous Cell Count (SUN scale), and:
   * are receiving no treatment; or
   * are receiving:

     * prednisone ≥ 10 mg/day (or equivalent dose of another corticosteroid), or
     * at least 1 systemic immunosuppressant other than corticosteroids, or
     * combination of prednisone ≥ 10 mg/day (or equivalent dose of another corticosteroid) and other systemic immunosuppressant.
   * Have inactive disease, defined as having 0.5+ Vitreous Haze or less and 0.5+ or less Vitreous Cell Count (SUN scale), and:
   * are receiving:

     * prednisone <10 mg/day (or equivalent dose of another corticosteroid), or
     * at least 1 systemic immunosuppressant other than corticosteroids, or
     * combination of prednisone <10 mg/day (or equivalent dose of another corticosteroid) and other systemic immunosuppressant.
   * Have posterior, intermediate, or panuveitis; for panuveitis, if an anterior component is present, it must be less than the posterior component.
   * Sufficient inflammation to require systemic treatment and, based on the Investigator's decision, warrants intravitreal treatment.
   * Best-corrected ETDRS visual acuity of 20/400 or better (approximately 20 letters) in the study eye.
   * Best-corrected ETDRS visual acuity of 20/400 or better in the fellow eye (approximately 20 letters).

Exclusion Criteria:

1. Patients with bilateral uveitis who are receiving systemic immunosuppressive therapy (e.g., methotrexate, cyclosporine, cyclophosphamide, chlorambucil, mycophenolate mofetil, tacrolimus, or azathioprine) other than prednisone or other corticosteroids for the treatment of uveitis and the uveitis in the fellow eye, in the opinion of the Investigator, cannot be controlled with standard local therapies alone;
2. Any significant ocular disease that could compromise the visual outcome in the study eye.
3. Intravitreal injections (including but not limited to anti-vascular endothelial growth factors 60 days prior to the baseline;
4. Posterior subtenon's or intravitreal injection of steroids 90 days prior to Baseline;
5. Intraocular surgery within 90 days prior to Day 0 in the study eye;
6. Capsulotomy within 30 days prior to Day 0 in the study eye;
7. History of vitreoretinal surgery or scleral buckling within 90 days prior to Day 0 in the study eye;
8. Any ocular surgery (including cataract extraction or capsulotomy) of the study eye anticipated within the first 180 days following Day 0;
9. Intraocular pressure ≥25 mmHg in the study eye (glaucoma patients maintained on no more than 2 topical medications with IOP <25 mmHg are allowed to participate);
10. Pupillary dilation inadequate for quality fundus photography in the study eye;
11. Media opacity that would limit clinical visualization, intravenous fluorescein angiography (IVFA), or OCT evaluation in the study eye;
12. Presence of any form of ocular malignancy in the study eye, including choroidal melanoma;
13. History of herpetic infection in the study eye or adnexa;
14. Presence of known active or inactive toxoplasmosis in either eye;
15. Ocular or periocular infection in either eye;
16. Participation in other investigational drug or device clinical trials within 30 days prior to Day 0, or planning to participate in other investigational drug or device clinical trials within 180 days following Day 0. This includes both ocular and non-ocular clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of uveitic attacks as assessed by vitreous haze and cells. | 6 months

SECONDARY OUTCOMES:
Incidence of adverse and serious adverse events | 6 months
  Incidence, frequencey, and severity of adverse events reported during the first 6 months of the study period.
Changes in central retinal thickness | 6 months
  Improvement or worsening of macular edema compared to baseline. Development of macular edema in patients with otherwise normal macualr thickness at baseline
Steroid sparing effect | 6 months
  Proportion of subjects with active uveitis who achieve complete or partial response to sirolimus at month 6 while discontinuing their steroid therapy.
  Proportion of subjects with inactive uveitis who maintain quiscent study eyes at month 6 while discontinuing their steroid therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Quan D Nguyen, MD, MSc, Principal Investigator — Stanford University Byers Eye Institute
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Derived] Teabagy S, Wood E, Bilsbury E, Doherty S, Janardhana P, Lee DJ. Ocular immunosuppressive microenvironment and novel drug delivery for control of uveitis. Adv Drug Deliv Rev. 2023 Jul;198:114869. doi: 10.1016/j.addr.2023.114869. Epub 2023 May 10. PMID 37172782